CLINICAL TRIAL: NCT05965271
Title: A Real World Study on Fabulous® Thoracic Aortic Stent System for Stanford B Aortic Dissection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Fabulous WQ-F02
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Aortic Dissection
Keywords: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fabulous Thoracic Aortic Stent System
  Interventions: Device: Fabulous Thoracic Aortic Stent System

INTERVENTIONS:
Device: Fabulous Thoracic Aortic Stent System — Endovascular treament in patients with aortic dissection with Fabulous Thoracic Aortic Stent System

SUMMARY:
A multicenter, retrospective study to evaluate the real-world efficacy of the Fabulous thoracic aortic stent system in the treatment of Stanford Type B aortic dissection.

DETAILED DESCRIPTION:
Fabulous Thoracic Aortic Stent System is specially designed for aortic dissection based on PETTICOAT technique.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old, regardless of gender;
* Subject was diagnosed with Stanford Type B dissection and treated with Fabulous thoracic aortic stent system, including either a covered stent system, a bare stent, or both;
* With appropriate arterial access and suitable for endovascular aortic repair;
* Subjects could understand the purpose of the trial, volunteered to participate in the study, signed the informed consent form by themselves or their legal representatives, and were willing to complete the follow-up as required by the protocol.

Exclusion Criteria:

* Patients have participated in clinical trials of other drugs or medical devices related to target lesion treatment or have participated in clinical trials of other drugs or medical devices and have not reached the primary endpoint;
* Patients were unable or unwilling to participate in the study;
* Patients were judged by the investigator to be ineligible for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stanford type B aortic dissection are treated with Fabulous Thoracic Aortic Stent System in the real world.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse events | within 30 days after operation
  Include all-cause death, aortic rupture, retrograde type A aortic dissection, distal stent graft induced new entry, endoleak, myocardial infarction, respiratory failure, renal failure, intestinal necrosis, permanent paraplegia, ischemic stroke, and severe lower limb ischemia.

SECONDARY OUTCOMES:
Immediate technical success | Immediate during operation
  Immediate technical success was defined as the stent was successfully delivered to the intended site and released.
Change of diameter | 30 days, 3 months,6 months after operation
  Changes of minimum diameter of true lumen, maximum diameter of false lumen and maximum total diameter of aorta before and after operation.
Major adverse events | 3 months,6 months after operation
  Include all-cause death, aortic rupture, retrograde type A aortic dissection, distal stent graft induced new entry, endoleak, myocardial infarction, respiratory failure, renal failure, intestinal necrosis, permanent paraplegia, ischemic stroke, and severe lower limb ischemia.
All-cause death and dissection related death | 3 months,6 months after operation
  All-cause deaths are defined as death from any cause during the follow-up. Dissection related death refers to death caused by rupture of aortic dissection or endovascular treatment of aortic dissection.
The incidence of reintervention | 30 days, 3 months,6 months after operation
  Thoracotomy or secondary intervention due to aortic dissection

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital Of Harbin Medical University, Harbin, Heilongjiang
  - Wuhan Asia General Hospital, Wuhan, Hubei
  - Central Hospital of Dalian University of Technology, Dalian, Liaoning
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Fu Weiguo, Shanghai
  - Shanghai Chest Hospital, Shanghai